CLINICAL TRIAL: NCT00005957
Title: A Phase III Study of Regional Radiation Therapy in Early Breast Cancer
Brief Title: Radiation Therapy in Treating Women Who Have Undergone Surgery for Early-Stage Invasive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NSABP Foundation Inc (Network); Radiation Therapy Oncology Group (Network); SWOG Cancer Research Network (Network); Trans Tasman Radiation Oncology Group (Other); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA20; CAN-NCIC-MA20; NSABP-CAN-NCIC-MA20 (Other: NSABP); NCCTG-CAN-NCIC-MA20 (Other: NCCTG); RTOG-CAN-NCIC-MA20 (Other: RTOG); SWOG-CAN-NCIC-MA20 (Other: SWOG); TROG-CAN-NCIC-MA20 (Other: TROG); CDR0000067938 (Other: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Breast Irradiation (Active Comparator)
  Interventions: Radiation: Standard Breast Irradiation
- Breast Radiation plus regional radiation (Experimental): regional radiation therapy (to the ipsilateral supraclavicular, axillary and internal mammary nodes)
  Interventions: Radiation: Breast Radiation plus Regional Radiation

INTERVENTIONS:
Radiation: Standard Breast Irradiation — Standard Breast Irradiation - A dose of 5000 cGy in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the standard tangent fields.
  Arms: Standard Breast Irradiation
Radiation: Breast Radiation plus Regional Radiation — Breast Radiation plus Regional Radiation - A dose of 5000 cGy in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the modified wide tangent fields.
  Arms: Breast Radiation plus regional radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiation to the tumor site and surrounding area may kill more tumor cells. It is not yet known if radiation therapy to the breast alone following surgery is more effective than radiation therapy to the breast plus surrounding tissue in treating invasive breast cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to the breast alone to see how well it works compared to radiation therapy to the breast plus surrounding tissue in treating women who have undergone surgery for early-stage invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival, disease-free survival, isolated local regional disease-free survival, and distant disease-free survival in women with previously resected, early stage, invasive breast cancer treated with breast radiotherapy with or without regional radiotherapy.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients (in certain participating centers) treated with these regimens.
* Compare the cosmetic outcomes in patients (in certain participating centers) treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of positive nodes (0 vs 1-3 vs more than 3), number of axillary nodes removed (<10, > or equal to 10); type of chemotherapy (anthracycline containing vs other vs none), hormonal therapy (yes vs no), number of axillary lymph nodes excised*, and participating center. Patients are randomized to one of two treatment arms.

NOTE: * Patients with a negative sentinel node dissection with or without an axillary dissection will be stratified according to the total number of nodes removed

* Arm I: Patients undergo standard breast radiotherapy alone 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo breast and regional radiotherapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.

Radiotherapy in both arms begins as soon as possible after randomization. Radiotherapy must begin within 8 weeks after completion of adjuvant IV chemotherapy, unless radiotherapy is administered concurrently with chemotherapy (i.e., cyclophosphamide, methotrexate, and fluorouracil [CMF]), or within 16 weeks after the last breast surgery for patients treated with hormonal therapy alone.

Quality of life is assessed (in patients in certain participating centers) within 2 weeks prior to randomization, during the last week of radiotherapy, at 3 and 9 months after completion of radiotherapy, and then annually until first distant disease recurrence.

Cosmetic outcome is assessed (in patients in certain participating centers) within 2 weeks prior to randomization, and then at 3 and 5 years after completion of radiotherapy or until first distant disease recurrence.

Patients are followed at 3, 6, and 9 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 1,822 patients will be accrued for this study within approximately 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven invasive carcinoma of the breast

  * No evidence of T4, N2-3, or M1 disease prior to surgery
  * Node positive or high-risk node negative
* Prior breast-conserving therapy (BCT) (e.g., lumpectomy, partial mastectomy, or segmental mastectomy) and axillary node dissection or sentinel node biopsy required and must be a candidate for breast radiotherapy after BCT

  * Normally patients should have microscopically clear resection margins and those with positive margins should undergo reexcision
  * Patients with microscopically focally positive margins (defined as no greater than 3 times high power fields) are candidates for breast radiotherapy plus a boost to the lumpectomy site
  * Patients with prior sentinel node dissection eligible if node negative, but still meet high-risk criteria

    * If node positive, then a level I and II axillary dissection must be performed
  * No evidence of residual disease in axilla after dissection
* Must be treated with currently accepted adjuvant systemic chemotherapy and/or hormonal therapy
* High risk of regional and systemic recurrence due to one of the following:

  * Pathologically positive axillary lymph nodes
  * Pathologically negative axillary lymph nodes with one of the following:

    * Primary tumor greater than 5 cm
    * Primary tumor greater than 2 cm and less than 10 axillary lymph nodes excised and one of the following:

      * Estrogen receptor negative
      * Skarf-Bloom-Richardson grade 3
      * Lymphovascular invasion
* Hormone receptor status:

  * Estrogen and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Sex:

* Female

Menopausal status:

* Premenopausal or postmenopausal

Performance status:

* ECOG 0-2

Life expectancy:

* At least 5 years

Hematopoietic:

* Not specified

Hepatic:

* SGOT and/or SGPT no greater than 3 times upper limit of normal (ULN)*
* Alkaline phosphatase no greater than 3 times ULN* NOTE: * Patients with laboratory values greater than 3 times ULN may still be eligible if no metastatic disease by imaging examinations

Renal:

* No serious nonmalignant renal disease

Cardiovascular:

* No serious nonmalignant cardiovascular disease

Pulmonary:

* No serious nonmalignant pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other serious nonmalignant disease (e.g., systemic lupus erythematosus or scleroderma) that would preclude definitive surgery or radiotherapy
* No other malignancy except:

  * Nonmelanomatous skin cancer
  * Carcinoma in situ of the cervix or endometrium
  * Contralateral noninvasive breast cancer (unless prior radiotherapy to the contralateral breast)
  * Invasive carcinoma of the cervix, endometrium, colon, thyroid, or melanoma that was curatively treated at least 5 years prior to study participation
* No psychiatric or addictive disorder that would preclude informed consent or study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Concurrent standard adjuvant chemotherapy allowed

Endocrine therapy:

* See Disease Characteristics
* Concurrent standard adjuvant hormonal therapy allowed

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Ages: 16 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1832 (Actual)
Dates: Start 2000-03-09 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Whelan, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; David S. Parda, Study Chair — Allegheny Cancer Center at Allegheny General Hospital; Julia R. White, MD, Study Chair — Medical College of Wisconsin; Lori J. Pierce, MD, Study Chair — University of Michigan Rogel Cancer Center; Boon Chua, MD, Study Chair — Peter MacCallum Cancer Centre, Australia; Laura A. Vallow, MD, Study Chair — Mayo Clinic
Locations (26):
- Canada (26):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Whelan TJ, Olivotto IA, Parulekar WR, Ackerman I, Chua BH, Nabid A, Vallis KA, White JR, Rousseau P, Fortin A, Pierce LJ, Manchul L, Chafe S, Nolan MC, Craighead P, Bowen J, McCready DR, Pritchard KI, Gelmon K, Murray Y, Chapman JA, Chen BE, Levine MN; MA.20 Study Investigators. Regional Nodal Irradiation in Early-Stage Breast Cancer. N Engl J Med. 2015 Jul 23;373(4):307-16. doi: 10.1056/NEJMoa1415340. PMID 26200977
- [Derived] Gross JP, Whelan TJ, Parulekar WR, Chen BE, Rademaker AW, Helenowski IB, Donnelly ED, Strauss JB. Development and Validation of a Nomogram to Predict Lymphedema After Axillary Surgery and Radiation Therapy in Women With Breast Cancer From the NCIC CTG MA.20 Randomized Trial. Int J Radiat Oncol Biol Phys. 2019 Sep 1;105(1):165-173. doi: 10.1016/j.ijrobp.2019.05.002. Epub 2019 May 11. PMID 31085285

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Breast Irradiation: radiation therapy: Standard Breast Irradiation - A dose of 5000 centigray (cGy) in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the standard tangent fields.
Period: Overall Study
Arm/Group | Standard Breast Irradiation | Breast Radiation Plus Regional Radiation
Started | 916 | 916
Completed | 908 | 888
Not Completed | 8 | 28
Not completed — No treated | 3 | 9
Not completed — Crossover to the other arm | 5 | 19

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Standard Breast Irradiation: radiation therapy: Standard Breast Irradiation - A dose of 5000 cGy in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the standard tangent fields.
- Total: Total of all reporting groups
Arm/Group | Standard Breast Irradiation | Breast Radiation Plus Regional Radiation | Total
Number analyzed (Participants) | 916 | 916 | 1832
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 54 (10) | 54 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 916 | 916 | 1832
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Duration of study
Time Frame: 10 years
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of alive at 10 years
Arm/Group | Standard Breast Irradiation | Breast Radiation Plus Regional Radiation
Number analyzed (Participants) | 916 | 916
percentage of alive at 10 years | 82 [79 to 84] | 83 [80 to 85]
Statistical Analysis 1: Comparison: Standard Breast Irradiation vs Breast Radiation Plus Regional Radiation; It was estimated that the actuarial five year survival of patients on the control arm of this trial would be 80% and a 5% increase in five year survival with experiment arm is clinically interesting to detect. A sample size of 1832 will ensure 80% power to detect such a difference with two-sided alpha of 0.05; Test type: Superiority or Other; p = 0.38, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.72 to 1.13] — Hazard ratio (HR) estimation is for Standard Breast Irradiation arm versus Breast Radiation plus regional radiation arm

2. Secondary Outcome: Disease-free Survival
Description: Disease-free survival (including locoregional and distant disease)
Time Frame: 10 years
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of disease-free at 10 years
Arm/Group | Standard Breast Irradiation | Breast Radiation Plus Regional Radiation
Number analyzed (Participants) | 916 | 916
percentage of disease-free at 10 years | 77 [74 to 80] | 82 [79 to 85]
Statistical Analysis 1: Comparison: Standard Breast Irradiation vs Breast Radiation Plus Regional Radiation; Test type: Superiority or Other; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.61 to 0.94]

ADVERSE EVENTS:
Time Frame: 10 years
Groups:
- Standard Breast Irradiation: radiation therapy: Standard Breast Irradiation - A dose of 5000 cGy in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the standard tangent fields.
  Analysis of adverse events were based on the 927 patients who actually received Standard Breast Irradiation treatment. A total of 908 patients who were randomized to Standard Breast Irradiation and 19 patients who were randomized to Breast Radiation plus regional radiation actually received the Standard Breast Irradiation treatment.
- Breast Radiation Plus Regional Radiation: regional radiation therapy (to the ipsilateral supraclavicular, axillary and internal mammary nodes)
  Breast Radiation plus Regional Radiation - A dose of 5000 cGy in 25 fractions at a rate of 200 cGy per day, 5 days a week for 5 weeks will be prescribed to the modified wide tangent fields.
  Analysis of adverse events were based on the 893 patients who actually received Breast Radiation plus regional radiation treatment. A total of 5 patients who were randomized to Standard Breast Irradiation and 888 patients who were randomized to Breast Radiation plus regional radiation actually received the Breast Radiation plus regional radiation treatment.
Arm/Group | Standard Breast Irradiation | Breast Radiation Plus Regional Radiation
Serious Adverse Events (participants affected / at risk) | 1/927 | 3/893
Other Adverse Events (participants affected / at risk) | 745/927 | 752/893
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Breast Irradiation (N=927) | Breast Radiation Plus Regional Radiation (N=893)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Breast Irradiation (N=927) | Breast Radiation Plus Regional Radiation (N=893)
Lymphedema (Blood and lymphatic system disorders) | 180 | 226
Fatigue (General disorders) | 353 | 343
Pain due to radiation (General disorders) | 252 | 233
Joint (General disorders) | 69 | 89
Skin (General disorders) | 313 | 316
Subcutaneous tissue (General disorders) | 167 | 180
Radiation dermatitis (Injury, poisoning and procedural complications) | 126 | 130
Muscle weakness (Musculoskeletal and connective tissue disorders) | 131 | 157
Myalgia (Musculoskeletal and connective tissue disorders) | 197 | 217
Neuropathy-sensory (Nervous system disorders) | 187 | 218
Neuropathic pain (Nervous system disorders) | 110 | 96
Gynecomastia (Reproductive system and breast disorders) | 283 | 256
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 116
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 118 | 150
Hot flashes/ flushes (Vascular disorders) | 65 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No